CLINICAL TRIAL: NCT07242092
Title: Effect of Methotrexate Discontinuation on Immunogenicity of 20-valent Pneumococcal Conjugate Vaccine (PCV20) in Patients With Autoimmune Rheumatic Diseases
Brief Title: Influence of Methotrexate Discontinuation on Immunogenicity After PCV-20 Vaccine in Patients ARDs
Acronym: MTX-PCV20-ARD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Insituto Adolfo Lutz (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 85236924.4.0000.0068
Record Dates: First submitted 2025-09-19; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Autoimmune Rheumatic Diseases
Keywords: Pneumococcal Vaccine; Methotrexate; PCV20; Immunogenicity; Vaccination; Rheumatology
MeSH Terms: interventions — Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTX suspension (Experimental): Participants randomized to this arm will receive one dose of the 20-valent pneumococcal conjugate vaccine (PCV20) at baseline (D0). They will be instructed to discontinue methotrexate (MTX) for 2 weeks following vaccination, then resume their regular MTX regimen. Prednisone up to 5 mg/day and other stable background therapies will be maintained. Blood samples will be collected at baseline (D0), 4 weeks post-vaccination (D28), and 6 months post-vaccination (D180).
  Interventions: Biological: Pneumococcal Vaccine
- MTX (Active Comparator): Participants randomized to this arm will receive one dose of the 20-valent pneumococcal conjugate vaccine (PCV20) at baseline (D0). They will continue MTX therapy without interruption during the vaccination period, maintaining their stable immunosuppressive regimen. Prednisone up to 5 mg/day and other stable background therapies will also be maintained. Blood samples will be collected at baseline (D0), 4 weeks post-vaccination (D28), and 6 months post-vaccination (D180).
  Interventions: Biological: Pneumococcal Vaccine

INTERVENTIONS:
Biological: Pneumococcal Vaccine — All participants will receive a single intramuscular dose (0.5 mL) of PCV20 (Prevnar 20®, Pfizer), administered into the deltoid muscle at baseline (Day 0). PCV20 contains purified capsular polysaccharides of 20 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F), individually conjugated to the nontoxic diphtheria CRM197 carrier protein. The conjugation induces a T-cell dependent immune response, resulting in higher-affinity antibodies and immune memory compared to polysaccharide vaccines.
  Other Names: 20-valent Pneumococcal Conjugate Vaccine (PCV20)

SUMMARY:
This clinical trial aims to evaluate the effect of temporary methotrexate (MTX) discontinuation on the humoral immunogenicity of the 20-valent pneumococcal conjugate vaccine (PCV20) in adult patients with autoimmune rheumatic diseases (ARDs).

Key questions:

* Does suspending MTX for 2 weeks after PCV20 enhance humoral immunogenicity?
* What is the impact of MTX discontinuation on functional opsonophagocytic activity (OPA) and cellular immunity?
* What is the risk of disease flaring with MTX withdrawal?

DETAILED DESCRIPTION:
Patients with autoimmune rheumatic diseases (ARDs) have an increased risk of infections, including invasive pneumococcal disease, due to underlying immune dysregulation and the frequent use of immunosuppressive therapies. Pneumococcal vaccination is strongly recommended in this population; however, methotrexate (MTX), a cornerstone therapy for ARDs, has been consistently associated with reduced vaccine immunogenicity.

Evidence from randomized clinical trials in influenza and COVID-19 vaccination has demonstrated that short-term MTX discontinuation (10-14 days post-vaccination) can significantly enhance humoral immune responses. However, this strategy may be accompanied by an increased risk of mild disease flare. Importantly, no study to date has evaluated the effect of temporary MTX discontinuation on pneumococcal vaccination, representing a critical knowledge gap in the care of immunosuppressed patients.

The 20-valent pneumococcal conjugate vaccine (PCV20) represents the most comprehensive pneumococcal conjugate vaccine currently licensed, covering 20 serotypes responsible for the majority of invasive disease. Unlike polysaccharide vaccines, conjugate vaccines generate T-cell dependent immune responses, leading to higher-quality and longer-lasting protection. Yet, the immunogenicity of PCV20 in patients with ARDs under MTX therapy has not been investigated.

This randomized, double-blind, controlled clinical trial will evaluate the impact of a 2-week MTX discontinuation following PCV20 vaccination in patients with ARDs in remission or low disease activity. A total of 192 adult patients will be enrolled and randomized 1:1 to either suspend MTX for 2 weeks after vaccination or continue MTX treatment as usual.

All participants will receive one dose of PCV20 at baseline (D0). Blood samples will be collected at baseline (D0), 4 weeks post-vaccination (D28), and 12 months post-vaccination (D180). Humoral immunogenicity will be assessed by quantifying IgG antibody concentrations against 12 vaccine serotypes using multiplex Luminex assays. In addition, we will evaluate serotype-specific opsonophagocytic activity (OPA) assays to assess functional antibody responses.

Disease activity will be monitored throughout the study using standardized indices (DAS28 for rheumatoid arthritis, ASDAS for spondyloarthritis, SLEDAI for systemic lupus erythematosus, MMT for myopathies, among others).

Safety assessments will include the recording of local and systemic adverse events in structured diaries and surveillance for disease flares, with predefined management protocols.

The primary endpoint is the seroconversion rate at 4 weeks after PCV20, defined as at least a twofold increase in IgG antibody levels for ≥50% of included serotypes.

Secondary endpoints include persistence of humoral immunity at 6 months, OPA titers, disease flare rates and adverse events.

By directly addressing the effect of MTX on PCV20 immunogenicity and incorporating both functional and cellular immune measures, this trial will generate critical evidence to guide vaccination strategies in immunosuppressed patients with ARDs and has the potential to inform future international guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>=18 years ) with confirmed ARD diagnosis (e.g., RA, PsA, axial SpA, primary Sjögren's, SLE, IIM, SSc, MCTD).
* Stable MTX dose ≥12 weeks.
* Prednisone ≤5 mg/day.
* Low disease activity/remission according to specific disease activity criteria.
* Eligible for PCV20 vaccination (no prior PCV20).

Exclusion Criteria:

* Anaphylaxis to vaccine components.
* Acute febrile illness.
* Guillain-Barré, decompensated CHF (NYHA III-IV), demyelinating disease.
* Live vaccine ≤4 weeks or inactivated vaccine ≤2 weeks before.
* Blood products in last 6 months.
* Severe infection in last month (including pneumococcal).
* Hospitalization at enrollment.
* Refusal to participate or inability to complete study procedures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion Rate After Vaccination | Day 28 (4 weeks post-vaccination).
  Proportion of participants who achieve seroconversion, defined as at least a twofold increase in IgG antibody concentrations for ≥50% of PCV20 vaccine serotypes (1, 3, 4, 5, 6B, 7F, 8, 9V, 14, 19F, 22F and 23F) compared to baseline, measured by multiplex Luminex assay.

SECONDARY OUTCOMES:
Opsonophagocytic Activity (OPA) Response | Day 0 to Day 28
  Functional antibody response will be assessed according to the serotype-specific opsonophagocytic activity (OPA), defined as at least a twofold increase in IgG antibody concentrations for ≥50% of vaccine serotypes (6B, 8, 14, 19A, 22F and 23F) compared to baseline.
Persistence of Humoral Immunity | Day 180 (6 months post-vaccination).
  Persistence of IgG antibody response assessed by Luminex and OPA assays by specific vaccine serotypes (1, 3, 4, 5, 6B, 7F, 8, 9V, 14, 19F, 22F and 23F).
Frequency of Disease Flares in Rheumatoid Arthritis | Baseline through Day 28.
  To assess the effect of temporary MTX discontinuation on disease activity in participants with rheumatoid arthritis, as measured by the Disease Activity Score 28 (DAS28). The DAS28 includes a count of tender and swollen joints (out of 28), a measure of general health (VAS), and either ESR or CRP. Scores range from approximately 0.9 to 9.4, with higher scores indicating worse disease activity.
Frequency of Disease Flares in Spondyloarthritis | Baseline through Day 28
  To evaluate the impact of MTX discontinuation on disease activity in participants with spondyloarthritis, as measured by the Ankylosing Spondylitis Disease Activity Score (ASDAS). The ASDAS combines patient-reported outcomes (back pain, duration of morning stiffness, peripheral pain/swelling, and global assessment) and an objective measure of inflammation (CRP or ESR). Scores range from approximately 0.6 to 6, with higher values indicating worse disease activity.
Frequency of Disease Flare in Systemic Lupus Erythematosus | Baseline through Day 28
  To assess the frequency of disease flares in participants with systemic lupus erythematosus following MTX discontinuation, using the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K). SLEDAI-2K scores range from 0 to 105, with higher scores indicating more severe disease activity. A flare is defined as an increase in SLEDAI-2K score from baseline based on pre-established thresholds.
Frequency of Disease Flare in Myopathies | Baseline through Day 28
  To evaluate the impact of MTX discontinuation on muscle strength in patients with idiopathic inflammatory myopathies, using the Manual Muscle Testing-8 (MMT-8) scale. The MMT-8 score ranges from 0 to 80, with higher scores indicating greater muscle strength and better clinical outcomes. A decrease in score indicates clinical worsening.
Frequency of Disease Flares in Psoriatic Arthritis | Baseline through Day 28
  To assess the frequency of disease flares following MTX discontinuation in participants with Psoriatic Arthritis, using the Disease Activity Index for Psoriatic Arthritis (DAPSA). Disease flares will be defined as worsening in disease activity classification (e.g., from remission to low, or from low to moderate activity). The DAPSA score ranges as follows: Remission (0-4), Low (5-14), Moderate (15-28) and High (>28). Higher scores indicate worse disease activity.
Frequency of Disease Flares in Primary Sjögren's Syndrome | Baseline through Day 28
  To evaluate the frequency of disease flares after MTX discontinuation in participants with primary Sjögren's Syndrome using the EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI). Disease flare will be defined as a clinically significant increase in ESSDAI score. The total ESSDAI score ranges from 0 to 123, with higher scores indicating more severe disease activity.
Frequency of Disease Flares in Behçet's Disease | Baseline through Day 28
  To determine the frequency of disease flares in patients with Behçet's Disease following MTX discontinuation, using the Behçet's Disease Current Activity Form - Simplified (BDCAF-s). Disease activity will be evaluated based on the presence and severity of clinical features (e.g., oral/genital ulcers, ocular involvement, skin lesions, etc.). Flare will be defined as the appearance or worsening of clinical manifestations as documented in the BDCAF-s.
Frequency of Disease Flares in Systemic Sclerosis | Baseline through Day 28
  To evaluate the frequency of disease flares in systemic sclerosis after MTX discontinuation using a composite clinical approach. Flare will be defined as the occurrence of one or more of the following:
  Increase in modified Rodnan Skin Score, Development of new digital ulcers, Worsening dyspnea score, Significant clinical change based on the EULAR disease activity assessment for systemic sclerosis.
Adverse events | Baseline through Day 28
  Safety will be closely monitored, and all serious adverse events will be classified as related or unrelated to the vaccine. A standardized adverse event diary will be provided to all patients and healthy controls for recording local and systemic reactions during the 4 weeks following each vaccine dose. Local reactions include: injection site pain, redness, swelling, bruising, itching, and induration. Systemic reactions include: fever, fatigue, chills, malaise, drowsiness, loss of appetite, nausea, vomiting, diarrhea, abdominal pain, dizziness, tremors, headache, fatigue, myalgia, muscle weakness, arthralgia, pruritus, and skin rash.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frenck RW Jr, Gurtman A, Rubino J, Smith W, van Cleeff M, Jayawardene D, Giardina PC, Emini EA, Gruber WC, Scott DA, Schmole-Thoma B. Randomized, controlled trial of a 13-valent pneumococcal conjugate vaccine administered concomitantly with an influenza vaccine in healthy adults. Clin Vaccine Immunol. 2012 Aug;19(8):1296-303. doi: 10.1128/CVI.00176-12. Epub 2012 Jun 27. PMID 22739693
- [Background] Chapman TJ, Pichichero ME, Kaur R. Comparison of pneumococcal conjugate vaccine (PCV-13) cellular immune responses after primary and booster doses of vaccine. Hum Vaccin Immunother. 2020 Dec 1;16(12):3201-3207. doi: 10.1080/21645515.2020.1753438. Epub 2020 May 13. PMID 32401658
- [Background] Ribeiro AC, Guedes LK, Moraes JC, Saad CG, Aikawa NE, Calich AL, Franca IL, Carvalho JF, Sampaio-Barros PD, Goncalves CR, Borba EF, Timenetsky Mdo C, Precioso AR, Duarte A, Bonfa E, Laurindo IM. Reduced seroprotection after pandemic H1N1 influenza adjuvant-free vaccination in patients with rheumatoid arthritis: implications for clinical practice. Ann Rheum Dis. 2011 Dec;70(12):2144-7. doi: 10.1136/ard.2011.152983. Epub 2011 Aug 22. PMID 21859696
- [Background] ten Wolde S, Breedveld FC, Hermans J, Vandenbroucke JP, van de Laar MA, Markusse HM, Janssen M, van den Brink HR, Dijkmans BA. Randomised placebo-controlled study of stopping second-line drugs in rheumatoid arthritis. Lancet. 1996 Feb 10;347(8998):347-52. doi: 10.1016/s0140-6736(96)90535-8. PMID 8598699